CLINICAL TRIAL: NCT03173352
Title: A Prospective Study on the Incidence and Related Risk Factors of Infantile Hemangioma in China
Acronym: IH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Yao Xiaojian, Principal Investigator, Zhujiang Hospital
Other Study IDs: Yao Xiaojian
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Infantile Hemangioma; Capillary Hemangioma; Capillary Hemangiomas; Hemangioma, Capillary Infantile; Strawberry Hemangioma
Keywords: Hemangioma
MeSH Terms: conditions — Hemangioma, Capillary; Hemangioma, capillary infantile; Hemangioma, Cavernous; Hemangioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infant hemangioma(IH): Infant hemangioma(IH) is the most common benign vascular tumor of infancy with the estimated incidence varies 1% to 12%.However, in China, the incidence of infant hemangioma and related epidemiological data remains unclear. So, We designed the study to collect data about both epidemiology related risk ractors of infantile hemangioma in China.

SUMMARY:
Infant hemangioma(IH) is the most common benign vascular tumor of infancy with the estimated incidence varies 1% to 12%.However, in China, the incidence of infant hemangioma and related epidemiological data remains unclear. So, the investigators designed the study for the following purposes: 1, to aware the incidence of infantile hemangioma and understand the related risk factorsin China; 2, to understand the clinical characteristics of infantile hemangioma and the risk factors for complications; 3, to investigate the level of knowledge, treatment options in infant hemangioma in Chinese doctors; 3, to improve the awareness of infantile hemangioma in parents and provide more advice for pregnancy counseling and eugenics.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* The infants within 12 months of age

Exclusion Criteria:

* Those whoes guardian does not want his data to be collected in this study

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants from the selected community
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of infantile hemangioma in China | about 1 years
  Data collected by questionnaire of infantile hemangioma, filled by the investigators

CONTACTS AND LOCATIONS:
Overall Officials: Tangde Zhang, Doctor, Study Director — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China